CLINICAL TRIAL: NCT04899609
Title: Behavioral Adaptation to Negative and Positive Social Signals in Healthy Volunteers
Brief Title: The Effects of Anger and Joy Expressions on Approach and Avoidance Behaviors in Healthy Volunteers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0304
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Episode
Keywords: Emotion; Motivation; Decision making; Goal-director behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Social interactions are part of our daily lives. Communicating with others is a recurring choice which is based on emotional cues, such as facial expression. Our action must be adapted to the emotional state of our interlocutor, otherwise the investigators will have poor quality interactions An emotional stimulus would cause a conditioned response (innate reaction). Thus, the presence of an angry person would automatically trigger flight behavior. More recently, however, it has been envisioned that this same avoidance behavior could be the result of a goal-directed behvior. In this case, the avoidance behavior would be the result of an evaluation of the consequences of the selected action. These goal-directed behaviors are guided by a mental representation of consequences The project aims to study behavioral choices (approach and avoidance) in response to negative and positive social cues (anger and joy) in 40 healthy volunteers using a computerized neuropsychological task, and to determine wheter these choices are the result of goal-directed behavior.

The study also aims to assess the modulation of behavioral adaptation by the level of impulsivity, lonilness, empathy, and by the capcity to understand others' intenstions.

ELIGIBILITY:
Inclusion criteria:

* Being between 18 and 65 years old
* Absence of psychiatric pathology over the entire life
* Being able to understand the nature, purpose and methodology of the study

Exclusion criteria:

* Mental retardation or sever medical co-morbidity
* Sensory or cognitive disability
* Pregnant or breastfeeding woman
* Protection by law (guardianship or curatorship)
* Deprivation of liberty (by judicial or administrative decision)
* Exclusion period in relation to another protocol
* Inability to understand, speak and write French

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of approach and avoidance behavior in response to positive (joy) and negative (anger) social signals | 1 day
  Calculation of the proportion of avoidance vs. approach choices

SECONDARY OUTCOMES:
Response time | 1 day
  Computerized measurement of reaction time before clicking to make the avoidance or approach choice

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Olie, MD PhD, Study Director — University Hospital, Montpellier
Locations (1):
- University hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC